CLINICAL TRIAL: NCT01789073
Title: Randomized, Controlled Trial Investigating the Effect of Preoperative Oral Immunonutrition on Complications and Length of Hospital Stay After Elective Surgery for Pancreatic Cancer
Brief Title: Preoperative Oral Immunonutrition for Patients With Pancreatic Cancer Undergoing Elective Surgery - Effect on Complications and Length of Hospital Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Arne Astrup, Chief of Institute of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-1-2012-146
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatic Cancer
Keywords: Postoperative; Complications; Elective; Surgery; GI surgery; Immunonutrition; Immune-enhancing; Immune-modulating; Nutrition; Pancreatic cancer; Postoperative complications and length of hospital stay after major gastrointestinal (GI) elective surgery.
MeSH Terms: conditions — Pancreatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Impact, Nestlé Health Science (Experimental): Oral Impact-arm receives the intervention the last 7 days prior to surgery
  Interventions: Dietary Supplement: Oral Impact, Nestlé Health Science
- Control (No Intervention): The control-arm receives no intervention but is treated according to the standard procedures

INTERVENTIONS:
Dietary Supplement: Oral Impact, Nestlé Health Science — Oral Impact from Nestlé Health Science. An enteral nutritional supplement high in protein and with added immune-enhancing nutrients: arginine, fish oil and nucleotides. The intervention arm receives Oral Impact in an individually estimated dosage according to a protein requirement of 1.5 g/kg bodyweight/day (subtracted their habitual protein intake). Each patient receives this dosage orally the last 7 days prior to surgery.
  Arms: Oral Impact, Nestlé Health Science

SUMMARY:
The purpose of this study is to investigate the effect of preoperative immunonutrition on complications and length of hospital stay in patients with pancreatic cancer undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women referred to treatment at Surgical Gastroenterology Clinic C, Ward 2122 for pancreatic cancer
* Age > 18 years.

Exclusion Criteria:

* Age < 18 years
* Pregnant and lactating women
* Persons who cannot understand and/or speak Danish
* Renal dysfunction
* Milk allergy
* Participants are excluded if elective surgery is not indicated after all

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall postoperative complications after major gastrointestinal (GI) elective surgery. | Within the first 30 days after surgery

SECONDARY OUTCOMES:
Length of hospital stay after major gastrointestinal (GI) elective surgery | Within the first 30 days after surgery

OTHER OUTCOMES:
Weight stability, functional capability and patients´ satisfaction with the overall study course. | from recruitment and within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Chief Phys., Ass. Prof., Principal Investigator — University of Copenhagen
Locations (1):
- Surgical Gastroenterology Clinic C, Ward 2122, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Gade J, Levring T, Hillingso J, Hansen CP, Andersen JR. The Effect of Preoperative Oral Immunonutrition on Complications and Length of Hospital Stay After Elective Surgery for Pancreatic Cancer--A Randomized Controlled Trial. Nutr Cancer. 2016;68(2):225-33. doi: 10.1080/01635581.2016.1142586. Epub 2016 Mar 4. PMID 26943500